CLINICAL TRIAL: NCT05899751
Title: High-dose Methotrexate Patterns of Use, Clearance, Toxicities, Supportive Care and Outcomes
Brief Title: Retrospective Registry Study of Patients With Cancer Treated With High-dose Methotrexate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Protherics Medicines Development Limited (Other)
Collaborators: Resonance Health (Industry)
Responsible Party: Sponsor
Organization: BTG International Inc. (Other)
Other Study IDs: PR001-CLN-pro101
Record Dates: First submitted 2023-04-11; First posted 2023-06-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-06

CONDITIONS: Acute Kidney Injury; Drug Toxicity
Keywords: Carboxypeptidases; Delayed Methotrexate Clearance; Hematologic Neoplasms; Hyperhydration; Leucovorin; Osteosarcoma
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions; Hematologic Neoplasms; Water Intoxication; Osteosarcoma | interventions — Methotrexate; glucarpidase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients Treated With High-dose Methotrexate: Patients with a diagnosis of any cancer receiving high-dose methotrexate chemotherapy.
  Interventions: Drug: High-dose methotrexate; Drug: Glucarpidase

INTERVENTIONS:
Drug: High-dose methotrexate — High-dose methotrexate
Drug: Glucarpidase — Glucarpidase

SUMMARY:
This retrospective observational study will evaluate high-dose methotrexate patterns of use, supportive care measures used during high-dose methotrexate chemotherapy, along with the incidence of delayed elimination of methotrexate, acute kidney injury and any associated impact of delayed elimination of methotrexate on future courses of chemotherapy and disease outcomes in adults and children with cancer.

The study will compare current practice with existing guidelines and best practices to identify potential gaps in the management of high-dose methotrexate administration and delayed elimination of methotrexate. The study will identify variations in practice and outcomes in different study centers, countries, cancer types, patient age groups, by different methotrexate doses and infusion times and different supportive care measures used. The study will also document the proportion of high-dose methotrexate courses in which glucarpidase has been used and any toxicities attributable to the use of glucarpidase.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of any cancer from January 1, 2001 to June 30, 2021.
* Receipt of high-dose methotrexate chemotherapy, defined as a dose of 500 mg/m2 of body surface area or higher.
* Medical records available for review.
* Any age; any cancer type.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at approximately 10 European sites where high-dose methotrexate infusions are administered. Sites will be selected to ensure a balanced accrual of children and adults treated with high-dose methotrexate.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Delayed Elimination of Methotrexate | 0-48 hours from the start of high-dose methotrexate infusion.
  Incidence of delayed elimination of methotrexate after high-dose methotrexate chemotherapy, defined by Ramsey criteria.
Acute Kidney Injury | 0-48 hours from the start of high-dose methotrexate infusion.
  Incidence of acute kidney injury of any grade after high-dose methotrexate chemotherapy.
Severe Delayed Elimination of Methotrexate | 0-48 hours from the start of high-dose methotrexate infusion.
  Incidence of severe delayed elimination of methotrexate after high-dose methotrexate chemotherapy, defined as a methotrexate level ≥2 standard deviations above the population mean at 36, 42, or 48 hours from the start of high-dose methotrexate infusion and with the presence of acute kidney injury of any grade.

SECONDARY OUTCOMES:
Severity of Acute Kidney Injury | 0-48 hours from the start of high-dose methotrexate infusion.
  Severity of occurrences of acute kidney injury using CTCAE v5 criteria.
Hospital Length of Stay | Assessed through study completion, up to 2 years after enrollment.
  Duration of hospitalization.
Hospital Readmission | Within 14 days of high-dose methotrexate infusion.
  Incidence of hospital readmission.
Delay of Subsequent Chemotherapy | Within 14 days of high-dose methotrexate infusion.
  Occurrence of delays to further blocks of chemotherapy resulting from delayed methotrexate elimination.
Dose Reduction or Omission of Subsequent High-dose Methotrexate Therapy | Within 14 days of high-dose methotrexate infusion.
  Occurrence of dose reduction or omission of high-dose methotrexate from further cycles of chemotherapy resulting from delayed methotrexate elimination.
Event-Free Survival | 3, 5, and 10 years.
  "Events" include death, relapse, abandonment, or refusal of treatment.
Overall Survival | 3, 5, and 10 years.
  All-cause mortality as well as mortality separately due to disease progression or toxicity.
Glucarpidase-Related Toxicity | 15 minutes post-glucarpidase through discharge.
  Occurrence of toxicities associated with glucarpidase, including frequency, severity (using CTCAE v5 criteria) and including documenting any toxicities of grade 3 or higher.
Methotrexate Clearance after Glucarpidase | 15 minutes post-glucarpidase through discharge.
  MTX levels.
Serum Creatinine Level | 15 minutes post-glucarpidase through discharge.
  Renal function, as measured by serum creatinine level.
Use of Subsequent High-Dose Methotrexate After Glucarpidase | Within 14 days of high-dose methotrexate infusion.
  Occurrence of subsequent high-dose methotrexate chemotherapy cycles given after glucarpidase.
Disease Outcome After Glucarpidase | 3, 5, and 10 years.
  Disease outcome after glucarpidase
Use of Hyperhydration | Assessed at time of hospital discharge.
  Incidence of the use of hyperhydration supportive care measures during high-dose methotrexate chemotherapy.
Use of Leucovorin | Assessed at time of hospital discharge.
  Incidence of the use of leucovorin during high-dose methotrexate chemotherapy.
Use of Dialysis or Hemofiltration | Assessed at time of hospital discharge.
  Incidence of the use of dialysis or hemofiltration during high-dose methotrexate chemotherapy.
Use of Oral Methotrexate Binders | Assessed at time of hospital discharge.
  Incidence of the use of oral methotrexate binders (cholestyramine, activated charcoal) during high-dose methotrexate chemotherapy.
Creatinine Clearance | 15 minutes post-glucarpidase through discharge.
  Renal function, as measured by creatinine estimate
Need for Dialysis | 15 minutes post-glucarpidase through discharge.
  Renal function, as measured by need for dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Rizzari, MD, Principal Investigator — University of Milano-Bicocca, Pediatric Hematology Oncology Unit MBBM Foundation
Locations (5):
- Assistance Publique Hôpitaux de Marseille (APHM), La Timone Hospital, Marseille, France
- University of Milan-Bicocca, Monza, Italy
- Spain (3):
  - Fundació Hospital Universitari Vall d'Hebron - Institut de Recerca (VHIR), Barcelona
  - Fundación Privada Instituto de Investigación Oncológica de Vall d'Hebron (VHIO), Barcelona
  - Hospital Universitario Reina Sofía, Córdoba

REFERENCES:
- [Background] Ramsey LB, Balis FM, O'Brien MM, Schmiegelow K, Pauley JL, Bleyer A, Widemann BC, Askenazi D, Bergeron S, Shirali A, Schwartz S, Vinks AA, Heldrup J. Consensus Guideline for Use of Glucarpidase in Patients with High-Dose Methotrexate Induced Acute Kidney Injury and Delayed Methotrexate Clearance. Oncologist. 2018 Jan;23(1):52-61. doi: 10.1634/theoncologist.2017-0243. Epub 2017 Oct 27. PMID 29079637
- [Background] Taylor ZL, Mizuno T, Punt NC, Baskaran B, Navarro Sainz A, Shuman W, Felicelli N, Vinks AA, Heldrup J, Ramsey LB. MTXPK.org: A Clinical Decision Support Tool Evaluating High-Dose Methotrexate Pharmacokinetics to Inform Post-Infusion Care and Use of Glucarpidase. Clin Pharmacol Ther. 2020 Sep;108(3):635-643. doi: 10.1002/cpt.1957. Epub 2020 Jul 18. PMID 32558929
- See also: A pharmacokinetic model for the dose of methotrexate to display the concentration vs time curve for an individual patient overlaid upon the population-predicted curve for that dose. — http://MTXPK.org
- See also: Voraxaze Summary of Product Characteristics (SmPC) — https://www.ema.europa.eu/en/documents/product-information/voraxaze-epar-product-information_en.pdf